CLINICAL TRIAL: NCT03983668
Title: Phase I/II Study of Pembrolizumab and In-situ Injection of CMP-001 in Patients With Relapsed and Refractory Lymphomas
Brief Title: CMP-001 for Relapsed and Refractory Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Umar Farooq (Other)
Collaborators: Checkmate Pharmaceuticals (Industry); Merck Sharp & Dohme LLC (Industry); University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Umar Farooq, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201902747
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CMP-001 plus pembrolizumab (Experimental): Intratumoral administration of CMP-001 and intravenous administration of pembrolizumab
  Interventions: Drug: CMP-001; Drug: Pembrolizumab

INTERVENTIONS:
Drug: CMP-001 — Immunostimulatory therapeutic agent
  Other Names: CYT003; QbG10; IND # 18627
Drug: Pembrolizumab — Humanized antibody used in cancer immunotherapy
  Other Names: Keytruda

SUMMARY:
This study is a single-arm, open-label, phase I/II trial designed to find a CMP-001 dose that, in combination with pembrolizumab, has optimal clinical efficacy and acceptable toxicity for patients with relapsed and refractory lymphomas.

DETAILED DESCRIPTION:
This is a single center, open-label, combined Phase I/II clinical study of intratumoral administration of CMP-001 and intravenous administration of pembrolizumab in selected participants with lymphoma. The key study objective is to find a CMP-001 dose that in combination with pembrolizumab has optimal clinical efficacy and acceptable toxicity. Dose-finding will be performed with an adaptive clinical trial design. Secondary study objectives include characterization of safety, pharmacodynamics, and assessment of anti-lymphoma activity.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically or cytologically confirmed diagnosis of relapsed or refractory Hodgkin Lymphoma or Non-Hodgkin Lymphoma (B and T cells).
* Male participants: A male participant must agree to use a contraception as detailed in Appendix C of this protocol during the treatment period and for at least five months after the final CMP-001 and pembrolizumab dose and refrain from donating sperm during this period.
* Female participants: A female participant is eligible to participate if she is not pregnant (see Appendix C), not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP) as defined in Appendix C OR
  2. A WOCBP who agrees to follow the contraceptive guidance in Appendix C during the treatment period and for at least 5 months after the last dose of study treatment.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial prior to the initiation of any study procedures. The participant must be capable of understanding and complying with protocol requirements.
* Have measurable disease based on Cheson 2007 (Cheson, et al 2007). Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Subjects must have at least one tumor lesion with a longest diameter of ≥ 1 cm that can be easily palpated or detected by ultrasound to facilitate intratumoral injection of CMP-001 (eg, tumor in skin, muscle, subcutaneous tissue or accessible lymph node).
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.
* Patients previously treated with anti B cell directed therapy, such as anti-B cell antibody therapy within the past year or a history of CAR T therapy at any time, will be evaluated for the presence of B cells by flow cytometry on peripheral blood. Patients with > 100 benign B cells will be considered eligible. Those with < 100 benign B cells may still be enrolled at the investigator's discretion but will only proceed to the therapeutic phase of the study if they have been shown to generate an anti-Qbeta antibody response, as demonstrated by ELISA assay, in response to the priming dose of vidutolimod

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to first dose of study drug. (see Appendix C). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137) within 4 weeks of enrollment into this trial.
* Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks or 5 half-lives whichever is shorter, prior to first dose of study drug.

Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with </= Grade 2 neuropathy may be eligible.

Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.

* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (</= 2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks or within 5 half-lives whichever is shorter, prior to the first dose of study treatment.

Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 2 weeks or within 5 half-lives whichever is shorter, after the last dose of the previous investigational agent.

* Has a diagnosis of primary immunodeficiency disorder or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (>/= Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patients with allotransplant in past 5 years or those with evidence of graft vs. host disease (GVHD) will be excluded.
* Have inadequate organ function as defined in the following table (Table 3). Specimens must be collected within 10 days prior to the start of study treatment.

  1. Hematological: Absolute neutrophil count (ANC) ≥1000/µL;Platelets ≥75 000/µL; Hemoglobin ≥8.0 g/dLa;
  2. Renal: Creatinine OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN;
  3. Hepatic: Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN; AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases);
  4. Coagulation: International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants;

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.

b Creatinine clearance (CrCl) should be calculated per institutional standard. Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | From the start of treatment up to two years
  To examine the toxicity related to the therapy by measuring the number of treatment related adverse events in patients
Objective response rate with statistical analysis based on the EffTox method | From the start of treatment up to two years
  The primary statistical analysis is based on the EffTox method of Thall and Cook (Thall and Cook 2004 [1], Thall, et al 2014 [2]). An adaptive escalation schema is used to find a dose with optimal clinical efficacy and acceptable toxicity. The design has a minimum sample size of 3 patients and a maximum of 39.

CONTACTS AND LOCATIONS:
Overall Officials: Umar Farooq, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thall PF, Cook JD. Dose-finding based on efficacy-toxicity trade-offs. Biometrics. 2004 Sep;60(3):684-93. doi: 10.1111/j.0006-341X.2004.00218.x. PMID 15339291
- [Background] Thall PF, Herrick RC, Nguyen HQ, Venier JJ, Norris JC. Effective sample size for computing prior hyperparameters in Bayesian phase I-II dose-finding. Clin Trials. 2014 Dec;11(6):657-66. doi: 10.1177/1740774514547397. Epub 2014 Sep 1. PMID 25179541